CLINICAL TRIAL: NCT00507572
Title: Collection of Outcomes Data for Pregnant Patients With Cancer
Status: Terminated | Type: Observational
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0518; NCI-2020-07509 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0518 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (medical chart review): Patients' medical records are reviewed prospectively and retrospectively.
  Interventions: Other: Medical Chart Review

INTERVENTIONS:
Other: Medical Chart Review — Medical records are reviewed
  Other Names: Chart Review

SUMMARY:
This study collects treatment and outcomes information on pregnant patients who are or were pregnant with cancer. Gathering and storing health information on pregnant patients with cancer, may provide data for future research studies and improve patient care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect, both prospectively and retrospectively, data on disease characterization, treatment and outcome for pregnant patients with malignancies seen at M. D. Anderson Cancer Center.

II. To organize clinical information in order to support multifaceted queries of patient characteristics, treatment, and pregnancy outcome data and to facilitate correlation of these characteristics with patient outcome.

III. To have a single data repository, kept on a secure platform, that will integrate clinical information and research findings and serve as a secure archive for future research.

OUTLINE:

Patients' medical records are reviewed prospectively and retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant patients with cancer and patients known to have been pregnant with a diagnosis of cancer are eligible, regardless of their diagnosis or treatment plan
* Patients may receive prenatal care from any obstetrician, but a consult with Maternal Fetal Medicine is encouraged

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients with cancer and patients known to have been pregnant with a diagnosis of cancer
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2005-12-19 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Creation of data repository for patient characteristics, treatment, and pregnancy outcome data | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Milbourne, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2005-12-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT00507572/ICF_000.pdf